CLINICAL TRIAL: NCT02702245
Title: Thylakoids' Effect on Glucose Homeostasis and Appetite Regulation After an Oral Glucose Tolerance Test in Healthy Volunteers
Brief Title: Effects of Two Doses of Thylakoids on OGTT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Eva-Lena Stenblom, M.D., Region Skane
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Thylakoid OGTT
Record Dates: First submitted 2016-02-25; First posted 2016-03-08 (Estimated); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Glucose Intolerance
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo comparator: Control (Placebo Comparator): OGTT without thylakoids.
  Interventions: Other: Placebo Comparator: Control
- Experimental: Thylakoids 5 g (Experimental): Intervention type: Dietary supplement. Supplement: thylakoid powder, dose 5 g. Intervention: OGTT at one occasion.
  Interventions: Dietary Supplement: Experimental: Thylakoids 5 g
- Experimental: Thylakoids 10 g (Experimental): Intervention type: Dietary supplement. Supplement: thylakoid powder, dose 10 g. Intervention: OGTT at one occasion.
  Interventions: Dietary Supplement: Experimental: Thylakoids 10 g

INTERVENTIONS:
Dietary Supplement: Experimental: Thylakoids 5 g — 75 g pure glucose + 5 g chloroplast membranes from spinach leaves in a dried powder.
  Other Names: Appethyl
  Arms: Experimental: Thylakoids 5 g
Dietary Supplement: Experimental: Thylakoids 10 g — 75 g pure glucose + 10 g chloroplast membranes from spinach leaves in a dried powder.
  Other Names: Appethyl
  Arms: Experimental: Thylakoids 10 g
Other: Placebo Comparator: Control — 75 g pure glucose.
  Arms: Placebo comparator: Control

SUMMARY:
This cross-over intervention study aims to investigate the effect of two doses of thylakoids to an oral glucose tolerance test (OGTT) on glucose and insulin homeostasis as well as appetite regulating hormones in healthy volunteers.

DETAILED DESCRIPTION:
A minimum of twenty healthy volunteers are recruited to participate in an OGTT at three different occasions separated by one week. At two of the occasions a green leaf extract, thylakoids, is added to a glucose solution; 5 gram or 10 gram in randomized order. The third occasion, without added thylakoids, serve as control.

Blood samples are taken fasting and 15, 30, 45, 60, 90, 120 and 180 minutes after the glucose load.

Blood samples are analysed for p-glucose, p-insulin, p-C-peptide, p-ghrelin, p-CCK and p-GLP-1.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Adult
* Normal-weight and weight stable
* Not pregnant or breast-feeding
* No use of medication that can affect glucose- and insulin homeostasis (for example corticosteroids).

Exclusion Criteria:

* Diabetes,
* Impaired glucose tolerance and/or insulin resistance
* Anaemia
* Use of tobacco or drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-01; Primary Completion 2016-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 180 minutes, repeated at three occasions
  Measurement of p-glucose, p-insulin and p-C-peptide in repeated blood sampling during three hours after an OGTT.

SECONDARY OUTCOMES:
p-GLP-1 | 180 minutes, repeated at three occasions
  Repeated blood sampling during three hours after an OGTT.
p-ghrelin | 180 minutes, repeated at three occasions
  Repeated blood sampling during three hours after an OGTT.

CONTACTS AND LOCATIONS:
Overall Officials: Eva-Lena Stenblom, M.D., Principal Investigator — Lund University, Region Skane

IPD SHARING:
Plan to Share IPD: No